CLINICAL TRIAL: NCT05419245
Title: Findings, Diagnostic Accuracy, Treatment, and Outcomes in Freeman-Burian Syndrome and Similar-appearing Arthrogryposis Syndromes: a Cross-sectional, Non-randomized Study
Brief Title: Survey Study and Records Review of Treatment Outcomes in Freeman-Sheldon Syndrome
Acronym: FINDFSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dufresne, Craig, MD, PC (Other)
Responsible Party: Sponsor
Other Study IDs: U1111-1120-5851
Record Dates: First submitted 2022-06-03; First posted 2022-06-15 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Freeman-Burian Syndrome; Freeman-Sheldon Syndrome; Whistling Face Syndrome; Sheldon-Hall Syndrome; Freeman-Sheldon Syndrome Variant; Arthrogryposis Distal Type 1; Arthrogryposis Distal Type 3; Gordon Syndrome
Keywords: craniofacial abnormalities; arthrogryposis; rehabilitation; surgery; therapy; health status; quality of life; patient reported outcome; health-related quality of life; depressive symptoms
MeSH Terms: conditions — Freeman-Sheldon syndrome; Distal arthrogryposis type 2B; Digitotalar Dysmorphism; Pseudohypoaldosteronism; Gordon syndrome; Craniofacial Abnormalities; Arthrogryposis; Depression | interventions — Multicenter Studies as Topic; Health Records, Personal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Freeman-Sheldon syndrome Classic Type: Patients who have all features required by the Stevenson criteria, including: very small mouth (microstomia); whistling-face appearance (pursed lips); "H" or "V" shaped chin dimple; very obvious down-slanting crease from the nostril to the corners of the mouth (nasolabial creases); and restricted movement in joints (contractures) of two or more body areas, often hands and feet, with fingers and toes frequently overlapping.
  Interventions: Other: Guided Health History for Freeman-Burian Syndrome Questionnaire; Other: Freeman-Burian syndrome Semi-Structured Quality of Life Interview; Other: Medical Records Review; Other: PTSD Checklist for DSM-5; Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale; Other: Review of Systems; Other: FACE-Q | Craniofacial - Appearance of the Face; Other: FACE-Q | Craniofacial - Appearance Distress; Other: FACE-Q | Craniofacial - Facial Function
- Freeman-Sheldon syndrome Craniofacial Type: Patients who have only the face and skull physical findings required by the Stevenson criteria, including: very small mouth (microstomia), whistling-face appearance (pursed lips), "H" or "V" shaped chin dimple, very obvious down-slanting crease from the nostril to the corners of the mouth (nasolabial creases).
  Interventions: Other: Guided Health History for Freeman-Burian Syndrome Questionnaire; Other: Freeman-Burian syndrome Semi-Structured Quality of Life Interview; Other: Medical Records Review; Other: PTSD Checklist for DSM-5; Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale; Other: Review of Systems; Other: FACE-Q | Craniofacial - Appearance of the Face; Other: FACE-Q | Craniofacial - Appearance Distress; Other: FACE-Q | Craniofacial - Facial Function
- Freeman-Sheldon syndrome Mixed Type: Patients who have the face and skull physical findings required by the Stevenson criteria and some but not all required joint problems.
  Interventions: Other: Guided Health History for Freeman-Burian Syndrome Questionnaire; Other: Freeman-Burian syndrome Semi-Structured Quality of Life Interview; Other: Medical Records Review; Other: PTSD Checklist for DSM-5; Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale; Other: Review of Systems; Other: FACE-Q | Craniofacial - Appearance of the Face; Other: FACE-Q | Craniofacial - Appearance Distress; Other: FACE-Q | Craniofacial - Facial Function
- Sheldon-Hall syndrome: Patients who have all features required by the Stevenson criteria, including: small mouth (not microstomia); neck webbing (pterygium colli); small but prominent chin; very obvious down-slanting crease from the nostril to the corners of the mouth (nasolabial creases); and restricted movement in joints (contractures) of two or more body areas, often hands and feet, with fingers and toes frequently overlapping.
  Interventions: Other: Guided Health History for Freeman-Burian Syndrome Questionnaire; Other: Freeman-Burian syndrome Semi-Structured Quality of Life Interview; Other: Medical Records Review; Other: PTSD Checklist for DSM-5; Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale; Other: Review of Systems; Other: FACE-Q | Craniofacial - Appearance of the Face; Other: FACE-Q | Craniofacial - Appearance Distress; Other: FACE-Q | Craniofacial - Facial Function
- Distal Arthrogryposis Type 1: Patients with features consistent with this diagnosis, including restricted movement in joints (contractures) of two or more body areas, often hands and feet, with fingers and toes frequently overlapping.
  Interventions: Other: Medical Records Review; Other: PTSD Checklist for DSM-5; Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale; Other: Review of Systems
- Distal Arthrogryposis Type 3: Patients with features consistent with this diagnosis, including: gap in the roof of the mouth (cleft palate); drooping eyelid (blepharoptosis); and spine curve problems; and restricted movement in joints (contractures) of two or more body areas, often hands and feet, with fingers and toes frequently overlapping.
  Interventions: Other: Medical Records Review; Other: PTSD Checklist for DSM-5; Other: Modified Flanagan Quality of Life Scale; Other: Center for Epidemiologic Studies Depression Scale; Other: Review of Systems; Other: FACE-Q | Craniofacial - Appearance of the Face; Other: FACE-Q | Craniofacial - Appearance Distress; Other: FACE-Q | Craniofacial - Facial Function

INTERVENTIONS:
Other: Guided Health History for Freeman-Burian Syndrome Questionnaire — Completed during the interview. The Guided Health History for Freeman-Burian Syndrome Questionnaire is a guided interview form that will be used to assess diagnosis, problems, treatments, and outcomes.
  Groups: Freeman-Sheldon syndrome Classic Type; Freeman-Sheldon syndrome Craniofacial Type; Freeman-Sheldon syndrome Mixed Type; Sheldon-Hall syndrome
Other: Freeman-Burian syndrome Semi-Structured Quality of Life Interview — Completed during the interview. Freeman-Burian syndrome Semi-Structured Quality of Life Interview is a quality of life interview for Freeman-Burian syndrome, taking into consideration individual's total health.
  Groups: Freeman-Sheldon syndrome Classic Type; Freeman-Sheldon syndrome Craniofacial Type; Freeman-Sheldon syndrome Mixed Type; Sheldon-Hall syndrome
Other: Medical Records Review — Review of medical records will be used, along with Guided Health History for Freeman-Burian Syndrome Questionnaire to assess patient histories and outcomes.
  Other Names: treatment records review; review of patient notes; patient chart review; review of clinical data
Other: PTSD Checklist for DSM-5 — Completed by patients before the interview. The PTSD Checklist for DSM-5 is a 20-item questionnaire. Each item is rated 0-4, with 0 being "Not at all" and 4 being "Extremely". Lower scores suggest the person may be experiencing fewer symptoms.
Other: Modified Flanagan Quality of Life Scale — Completed by patients before the interview. The Modified Flanagan Quality of Life Scale is a 16-item survey designed for use in persons with chronic illness. Each item is rated 1-7, with 1 being "Terrible" and 7 being "Delighted". Higher scores suggest the person may be experiencing a better quality of life.
Other: Center for Epidemiologic Studies Depression Scale — Completed by patients before the interview. The Center for Epidemiologic Studies Depression Scale is a 20-item survey that asks about depressive feelings and behaviours in the past week. Each item is rated 0-3, with 0 being "Rarely or none of the time (less than 1 day)" and 3 being "Most or all of the time (5-7 days)". Lower scores suggest the person may be experiencing fewer symptoms.
Other: Review of Systems — Completed during the interview. A review of systems is a checklist of medical problems.
  Other Names: health history; medical history
Other: FACE-Q | Craniofacial - Appearance of the Face — Completed by patients. The FACE-Q | Craniofacial - Appearance of the Face is a 9-item questionnaire. Each item is rated 1-4, with 1 being "Not at All" and 4 being "Very Much". Lower scores suggest the person may be less pleased with the appearance of their face.
  Groups: Distal Arthrogryposis Type 3; Freeman-Sheldon syndrome Classic Type; Freeman-Sheldon syndrome Craniofacial Type; Freeman-Sheldon syndrome Mixed Type; Sheldon-Hall syndrome
Other: FACE-Q | Craniofacial - Appearance Distress — Completed by patients. The FACE-Q | Craniofacial - Appearance Distress is an 8-item questionnaire. Each item is rated 1-4, with 1 being "Always" and 4 being "Never". Lower scores suggest the person may be experiencing more distress related to the appearance of their face.
  Groups: Distal Arthrogryposis Type 3; Freeman-Sheldon syndrome Classic Type; Freeman-Sheldon syndrome Craniofacial Type; Freeman-Sheldon syndrome Mixed Type; Sheldon-Hall syndrome
Other: FACE-Q | Craniofacial - Facial Function — Completed by patients. The FACE-Q | Craniofacial - Facial Function is a 10-item questionnaire. Each item is rated 1-3, with 1 being "I cannot do this" and 3 being "I can do this". Lower scores suggest the person may be experiencing more problems with facial muscle functioning.
  Groups: Distal Arthrogryposis Type 3; Freeman-Sheldon syndrome Classic Type; Freeman-Sheldon syndrome Craniofacial Type; Freeman-Sheldon syndrome Mixed Type; Sheldon-Hall syndrome

SUMMARY:
The purpose of this study is to evaluate the difference in diagnosis accuracy, treatment outcomes, patient perspectives, facial function and walking ability, emotional and social health, and respiratory complications between Freeman-Burian syndrome (formerly, Freeman-Sheldon or whistling face syndrome), Sheldon-Hall syndrome, and distal arthrogryposis types 3, and 1.

The approximate cumulative total time for study-related activities will be 3 hours, including email communication, survey completion, and a medical interview.

The study will involve completing 6 short ½ to 1-page surveys and participating in a medical interview. Participants may be asked to provide medical records for review. All study-related activities will take place remotely, and no travel is required.

DETAILED DESCRIPTION:
According to the only study of patients and a recent study of individual case reports, Freeman-Burian syndrome (FBS) may be over-diagnosed by 33-66%, and it is most often confused with Sheldon-Hall syndrome and distal arthrogryposis (DA) types 3 and 1. Unfortunately, while these conditions are different from FBS, many think of them as being less severe versions of FBS. This is not true. FBS is a skull and face syndrome, while Sheldon-Hall syndrome and DA types 1 and 3 are syndromes of the arms, legs, hands, and feet that (except DA type 1) may have mild face deformities. It is important to understand this difference, FBS does not respond well to treatment. The other syndromes generally do respond well to treatment. To improve diagnosis and treatment, it is important to understand factors contributing to an accurate diagnosis and treatment outcome. To provide better evidence for these being very different syndromes, it also is important to compare the above areas of health between people with all of these syndromes. It is hoped the study will help improve treatment and identify areas for further research.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are able to provide informed consent or have a legally appointed representative who is able to provide informed consent
* Patients who have Freeman-Burian syndrome (formerly, Freeman-Sheldon syndrome), Sheldon-Hall syndrome, distal arthrogryposis type 1, or distal arthrogryposis type 3
* Persons who speak and read English, German, Russian, or Czech

Exclusion Criteria:

* Patients who are not able to provide informed consent or do not have a legally appointed representative who is able to provide informed consent
* Patients who do not have Freeman-Burian syndrome (formerly, Freeman-Sheldon syndrome), Sheldon-Hall syndrome, distal arthrogryposis type 1, or distal arthrogryposis type 3
* Persons who do not speak or read English, German, Russian, or Czech

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: There are no patient enrollment restrictions based on gender, ethnicity, religion, socio-economic status, geographical location, or clinical setting.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Difference in intervention-related outcome rates between groups | During a single study interview, which lasts 1-2 hours
  Outcomes for all interventions are rated as either acceptable, unacceptable, or potentially harmful/harmful. Information related to outcomes of interventions is collected using the Guided Health History for Freeman-Burian Syndrome Questionnaire, Review of Systems forms, and Medical Records Review.
Difference in diagnostic accuracy between groups | During a single study interview, which lasts 1-2 hours
  This is the percent of patients with a stated diagnosis re-screened by study investigators with the same diagnosis. Diagnostic information is collected using the Guided Health History for Freeman-Burian Syndrome Questionnaire and Medical Records Review.

SECONDARY OUTCOMES:
Difference in posttraumatic stress disorder symptoms between groups | 1 week to 1 day before a single study interview, which lasts 1-2 hours
  Posttraumatic stress symptoms are assessed using the self-completed and validated PTSD Checklist for DSM-5, a 20-item questionnaire; each item is rated 0-4, with 0 being "Not at all" and 4 being "Extremely".
Difference in depressive symptoms between groups | 1 week to 1 day before a single study interview, which lasts 1-2 hours
  Depressive symptoms are assessed using the self-completed and validated Center for Epidemiologic Studies Depression Scale.
Difference in quality-of-life between groups | 1 week to 1 day before a single study interview, which lasts 1-2 hours
  Quality-of-life is scored using the self-completed Modified Flanagan Quality of Life Scale.
Difference in facial appearance satisfaction between groups | 1 week to 1 day before a single study interview, which lasts 1-2 hours
  Facial appearance satisfaction is scored using the self-completed FACE-Q | Craniofacial - Appearance of the Face.
Difference in facial appearance distress between groups | 1 week to 1 day before a single study interview, which lasts 1-2 hours
  Facial appearance distress is scored using the self-completed FACE-Q | Craniofacial - Appearance Distress.
Difference in facial muscle functioning symptoms between groups | 1 week to 1 day before a single study interview, which lasts 1-2 hours
  Facial muscle functioning symptoms are scored using the self-completed FACE-Q | Craniofacial - Facial Function.

OTHER OUTCOMES:
Difference in diagnostic accuracy between specialities between all sub-types of Freeman-Burian syndrome and the other diagnosis groups (Sheldon-Hall syndrome, distal arthrogryposis type 3, and distal arthrogryposis type 1) | During a single study interview, which lasts 1-2 hours
  Diagnostic accuracy is the percent of patients with a stated diagnosis re-screened by study investigators with the same diagnosis. Specialities include: orthopedics, plastic surgery, anesthesia, pediatrics, and medical genetics. Diagnostic information is collected using the Guided Health History for Freeman-Burian Syndrome Questionnaire and Medical Records Review.
Difference in head and face (craniofacial) surgery-related outcome rates between groups | During a single study interview, which lasts 1-2 hours
  Outcomes for all head and face (craniofacial) surgeries are rated as either acceptable, unacceptable, or harmful/potentially harmful. Information related to outcomes of interventions is collected using the Guided Health History for Freeman-Burian Syndrome Questionnaire, Review of Systems forms, and Medical Records Review.
Difference in spine surgery-related outcome rates between groups | During a single study interview, which lasts 1-2 hours
  Outcomes for all spine surgeries are rated as either acceptable, unacceptable, or harmful/potentially harmful. Information related to outcomes of interventions is collected using the Guided Health History for Freeman-Burian Syndrome Questionnaire, Review of Systems forms, and Medical Records Review.
Difference in foot and ankle surgery-related outcome rates between groups | During a single study interview, which lasts 1-2 hours
  Outcomes for all foot and ankle surgeries are rated as either acceptable, unacceptable, or harmful/potentially harmful. Information related to outcomes of interventions is collected using the Guided Health History for Freeman-Burian Syndrome Questionnaire, Review of Systems forms, and Medical Records Review.
Difference in hand and wrist surgery-related outcome rates between groups | During a single study interview, which lasts 1-2 hours
  Outcomes for all hand and wrist surgeries are rated as either acceptable, unacceptable, or harmful/potentially harmful. Information related to outcomes of interventions is collected using the Guided Health History for Freeman-Burian Syndrome Questionnaire, Review of Systems forms, and Medical Records Review.
Difference in other bone and joint surgery-related outcome rates between groups | During a single study interview, which lasts 1-2 hours
  Outcomes for other bone and joint surgeries are rated as either acceptable, unacceptable, or harmful/potentially harmful. Information related to outcomes of interventions is collected using the Guided Health History for Freeman-Burian Syndrome Questionnaire, Review of Systems forms, and Medical Records Review.
Difference in general anesthesia-related complication rates between groups | During a single study interview, which lasts 1-2 hours
  The course of general anesthesia-related is rated as either routine, minor, complication, major complication, or failure. Information related to complications of interventions is collected using the Guided Health History for Freeman-Burian Syndrome Questionnaire, Review of Systems forms, and Medical Records Review.
Difference in respiratory-related complication rates between groups | During a single study interview, which lasts 1-2 hours
  Respiratory-related complications are assessed using the Guided Health History for Freeman-Burian Syndrome Questionnaire. Additional information on physical findings is collected using the Review of Systems forms and from the Medical Records Review.
Difference in rates of difficulty eating (chewing and swallowing) between groups | During a single study interview, which lasts 1-2 hours
  Difficulty eating (chewing and swallowing) is assessed using the Guided Health History for Freeman-Burian Syndrome Questionnaire. Additional information on physical findings is collected using the Review of Systems forms and from the Medical Records Review.
Difference in rates of difficulty walking between groups | During a single study interview, which lasts 1-2 hours
  Difficulty walking is assessed using the Guided Health History for Freeman-Burian Syndrome Questionnaire. Additional information on physical findings is collected using the Review of Systems forms and from the Medical Records Review.
Qualitative difference in quality of life between groups | During a single study interview, which lasts 1-2 hours
  Qualitative assessment is done using the Freeman-Burian syndrome Semi-Structured Quality of Life Interview, a guided interview consisting of open-ended questions.

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Dufresne, MD, Principal Investigator — Dr Craig R Dufresne, MD, PC
Locations (1):
- Office of Craig R Dufresne, MD, PC, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be made available to other researchers.

REFERENCES:
- [Background] Poling MI, Dufresne CR, Chamberlain RL. Dr Ben Franklin and an unusual modern-day cure for recurrent pleuritis. Br J Gen Pract. 2017 Jan;67(654):32-33. doi: 10.3399/bjgp17X688705. No abstract available. PMID 28034943
- [Background] Poling MI, Dufresne CR. Head First, Not Feet First: Freeman-Sheldon Syndrome as Primarily a Craniofacial Condition. Cleft Palate Craniofac J. 2018 May;55(5):787-788. doi: 10.1177/1055665617753482. Epub 2018 Jan 25. PMID 29370530
- [Background] Poling MI, Dufresne CR. Revisiting the Many Names of Freeman-Sheldon Syndrome. J Craniofac Surg. 2018 Nov;29(8):2176-2178. doi: 10.1097/SCS.0000000000004802. PMID 30400128
- [Background] Poling MI, Dufresne CR, Chamberlain RL. Freeman-Burian syndrome. Orphanet J Rare Dis. 2019 Jan 10;14(1):14. doi: 10.1186/s13023-018-0984-2. PMID 30630514
- [Background] Poling MI, Dufresne CR. Epidemiology, prevention, diagnosis, treatment, and outcomes for psychosocial problems in patients and families affected by non-intellectually impairing craniofacial malformation conditions: a systematic review protocol of qualitative data. Syst Rev. 2019 May 27;8(1):127. doi: 10.1186/s13643-019-1045-1. PMID 31133050
- [Background] Poling MI, Dufresne CR. Freeman-Burian syndrome. Anasthesiologie und Intensivmedizin. 2019; 60(1): S8-S17. doi: 10.19224/ai2019.S008
- [Background] Poling MI, Dufresne CR, Portillo AL. Identification and Recent Approaches for Evaluation, Operative Counseling, and Management in Patients With Freeman-Burian Syndrome: Principles for Global Treatment. J Craniofac Surg. 2019 Nov-Dec;30(8):2502-2508. doi: 10.1097/SCS.0000000000005968. PMID 31567769
- [Background] Poling MI, Dufresne CR. Distal arthrogryposis type 3. Anasthesiologie und Intensivmedizin. 2019; 60(13): S536-S543. doi: 10.19224/ai2019.s536.
- [Background] Poling MI, Dufresne CR. Identification and Recent Approaches for Evaluation and Management of Dentofacial and Otolaryngologic Concerns for Patients With Freeman-Burian Syndrome: Principles for Global Treatment. J Craniofac Surg. 2020 May/Jun;31(3):787-790. doi: 10.1097/SCS.0000000000006155. PMID 31985597
- [Background] Poling MI, Dufresne CR, Chamberlain RL. Findings, Phenotypes, Diagnostic Accuracy, and Treatment in Freeman-Burian Syndrome. J Craniofac Surg. 2020 Jun;31(4):1063-1069. doi: 10.1097/SCS.0000000000006299. PMID 32149971
- [Background] Poling MI, Dufresne CR, McCormick RJ. Identification and Recent Approaches for Evaluation and Management of Rehabilitation Concerns for Patients with Freeman-Burian Syndrome: Principles for Global Treatment. J Pediatr Genet. 2020 Sep;9(3):158-163. doi: 10.1055/s-0040-1710339. Epub 2020 May 7. PMID 32714615
- [Background] Poling MI, Dufresne CR. Letter. AANA Journal. 2020; 88(5): 54.
- [Background] Poling MI, Dufresne CR. Letter: Precise Pulmonary Function Evaluation and Management of a Patient With Freeman-Sheldon Syndrome Associated With Recurrent Pneumonia and Chronic Respiratory Insufficiency (Ann Rehabil Med 2020;44:165-70). Ann Rehabil Med. 2020 Oct;44(5):409-410. doi: 10.5535/arm.20110. Epub 2020 Oct 29. No abstract available. PMID 33152847
- [Background] Poling MI, Dufresne CR. Accuracy of facts about Freeman-Sheldon syndrome. Clinical and Experimental Obstetrics and Gynecolology. 2021; 48(5): 997-998. doi: 10.31083/j.ceog4805160
- [Background] Poling MI, Dufresne CR. Diagnosis, evaluation, and treatment in Freeman-Burian syndrome: clinical practice guideline for a rare and complex craniofacial syndrome. Craniomaxillofacial Abstracts Presented at 78th Annual Meeting of the American Cleft Palate Craniofacial Meeting. FACE. 2021; 2(4): NP3. doi: 10.1177/27325016211049488
- [Background] Poling MI, Dufresne CR. Clarity on Diagnosis in Freeman-Burian syndrome. Turkiye Klinikleri Journal of Case Reports. doi: 10.5336/caserep.2022-88270 [In Press] Available online: 17 February 2022. Available at: https://www.turkiyeklinikleri.com/inpress_article/en-clarity-on-diagnosis-in-freeman-burian-syndrome-97915.html
- [Background] Poling MI, Dufresne CR. Oculoplastic surgery, diagnosis, and other matters in Freeman-Burian syndrome. Ophthalmic Genet. 2022 Jun;43(3):431-432. doi: 10.1080/13816810.2022.2068043. Epub 2022 Apr 28. No abstract available. PMID 35484845
- [Background] Poling MI, Dufresne CR. Anaesthesia recommendations for Sheldon-Hall syndrome. OrphanAnesthesia. 20 Feb 2019. Available at: https://www.orphananesthesia.eu/en/rare-diseases/published-guidelines/cat_view/61-rare-diseases/60-published-guidelines/237-sheldon-hall-syndrome.html
- [Background] Poling MI, Dufresne CR. Obstetrics and Diagnosis in Freeman-Burian syndrome. Version: 1. Authorea [preprint]. January 31, 2022. doi: 10.22541/au.164366820.09260728/v1.
- [Background] Poling MI, Dufresne CR. Misinformation and Misdiagnosis in Freeman-Burian syndrome. Version: 1. Authorea [preprint]. January 31, 2022. doi: 10.22541/au.164366815.52860865/v1.
- [Background] Poling MI, Dufresne CR. Limb Deformity Treatment and Diagnosis in Freeman-Burian syndrome. Version: 1. Authorea [preprint]. January 31, 2022. doi: 10.22541/au.164366820.05370920/v1.
- [Background] Poling MI, Dufresne CR. Unsafe Care and Misunderstanding Diagnosis in Freeman-Burian syndrome: Problems in Writing Case Reports Involving Rare Conditions and Strategies for Improvement. Authorea. January 24, 2022. doi: 10.22541/au.164303994.43963430/v1.
- [Background] Poling MI, Morales Corado JA, Chamberlain RL. Findings, phenotypes, and outcomes in Freeman-Sheldon and Sheldon-Hall syndromes and distal arthrogryposis types 1 and 3: protocol for systematic review and patient-level data meta-analysis. Syst Rev. 2017 Mar 6;6(1):46. doi: 10.1186/s13643-017-0444-4. PMID 28264711
- [Background] Poling MI, Dufresne CR. Re: "Periocular Anomalies in Freeman-Sheldon Syndrome". Ophthalmic Plast Reconstr Surg. 2022 Nov-Dec 01;38(6):609-610. doi: 10.1097/IOP.0000000000002307. Epub 2021 Nov 4. No abstract available. PMID 36326430
- See also: Principal Investigator's (Dr Craig R Dufresne) Research and Press Relations main webpage. Last Accessed: 7 Jun 2022 — https://www.duplastics.com/research-press/
- See also: "Freeman-Sheldon Syndrome" from the National Organization for Rare Disorders. Last Accessed: 10 Sept 2021 — https://rarediseases.org/rare-diseases/freeman-sheldon-syndrome/
- See also: Video about Freeman-Burian syndrome (previously known as Freeman-Sheldon syndrome) hosted by Genetic Alliance and presented by the Principal Investigator and Sub-Investigator (Craig R Dufresne and MI Poling). Last Accessed: 7 Jun 2022 — https://youtu.be/I3lTGDCl0Zk